CLINICAL TRIAL: NCT02500134
Title: Using AS-OCT to Assess the Role of Age and Region in the Morphology and Epithelial Thickness of Limbus
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201406106RINC
Record Dates: First submitted 2014-08-07; First posted 2015-07-16 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Limbus Corneae

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Normal: Healthy volunteer control without ocular surface disease or prior ophthalmic surgery history
  Interventions: Other: Optical coherence tomography study on limbus

INTERVENTIONS:
Other: Optical coherence tomography study on limbus — Optical coherence tomography study on limbus

SUMMARY:
The limbus located between the cornea and the conjunctiva tissue, is important for not only providing a barrier frontier to prevent conjunctival tissue invasion into the cornea, containing nerves passing to the cornea, having blood and lymph vasculature for oxygen and nutrient delivery, but also the niche environment of limbal stem cells.

So far, in vivo image systems are not able to visualize or identify the limbal stem cells directly. One alternative practical is to visualize the histological morphology of palisades of Vogt (POV), and to speculate the possible status of the stem cells accordingly. Slit-lamp biomicroscope can be used routinely for clinical examination of the limbal morphology. However, this technology does not allow for high resolution imaging of structural details and only up to 20% of patients can be identified. In vivo confocal microscopy has been used to visualize the POV and can provide cellular level resolution images, but the technique is limited by high magnification that restricts the area of the scan, and requires contact with the eye. Besides, both slit lamp biomicroscopy and in vivo confocal microscopy have the limitation of not being able to give an overall view of the dimension and structure of the whole palisades region.

Anterior segment optical coherence tomography (AS-OCT) is a noninvasive, rapid and reproducible technique to evaluate the anterior segment and can also provide in vivo spatial information. The purpose of the study is to assess the role of aging and regions on the limbus.

DETAILED DESCRIPTION:
The limbus located between the cornea and the conjunctiva tissue, approximately 1.5 mm wide in adult human eyes, is important for not only providing a barrier frontier to prevent conjunctival tissue invasion into the cornea, containing nerves passing to the cornea, having blood and lymph vasculature for oxygen and nutrient delivery, but also the niche environment of limbal stem cells. The human limbus contains radially oriented fibrovascular rides named palisades of Vogt (POV), a unique tissue first noted in 1866 and were further described in detail in 1921. The POV has unique structure, configuration and dimension which was commonly found in all types of epithelial stem cell niche all over the body, which include the complicated niche area providing a safe place to protect the stem cells from damage or injury. During the past few years, progress in stem cell research and cell therapy has focused attention on the POV as the location of the stem cells that keep the corneal epithelial homeostasis and clarity. The POV also provide the niche environment for limbal stem cells. The niche cells surrounding the limbal stem cells, the stromal environment underneath the limbal epithelial cells, the blood vessels and nerve innervation around the limbal epithelium all help create the unique niche environment for limabl stem cells. Understanding the limbal structure, especially the POV, is necessary for the treatment of limbal damage and the development of stem cell therapies targeted at restoring impaired function of limbal stem cells.

So far, in vivo image systems are not able to visualize or identify the limbal stem cells directly. One alternative practical is to visualize the histological morphology of POV, and to speculate the possible status of the stem cells accordingly. However, the microstructure of POV is not well defined or understood in spite of awareness of it's importance. Slit-lamp biomicroscope can be used routinely for clinical examination of the limbal morphology. However, this technology does not allow for high resolution imaging of structural details and only up to 20% of patients can be identified. In vivo confocal microscopy has been used to visualize the POV and can provide cellular level resolution images, but the technique is limited by high magnification that restricts the area of the scan. In addition, in vivo confocal microscopy requires direct contact with the eye. Although the quality of these images is impressive, the disadvantages existed included the direct contact during examination, the small field of view (~200μm x 200μm), and the limited axial resolution. Besides, both slit lamp biomicroscopy and in vivo confocal microscopy have the limitation of not being able to give an overall view of the dimension and structure of the whole palisades region.

Optical coherence tomography (OCT) is an imaging modality that allows for non-invasive imaging of the morphology of biological tissue with micrometer scale resolution at imaging depths of 1-2mm below the tissue surface. During these few years, OCT has become a useful clinical and research tool for imaging of the ocular surface. In addition to the mostly used application for observing the optic disc and retinal choroidial structure, the usage in the anterior segment, especially cornea, was also widely developed. An anterior segment OCT (Visante; Carl Zeiss Meditec, Dublin, CA), a time-domain OCT, is a commercial available OCT designed for especially for anterior segment. This OCT instrument has been used widely in LASIK, different lamellar keratoplasties, keratoconus screening and evaluation of corneal diseases in different layers. However, its limited resolution does not allow for the observation of the epithelial layer on the ocular surface. Spectral domain OCT with a corneal module can provide much better resolution than time domain OCT for the observation of epithelial layer on ocular surface. It has been used recently to evaluate the corneal epithelial layer with reliable results. In this study, we use a fourier-domain optical coherence tomography OCT (RTvue, Optovue Inc., Fremont, CA), with a corneal-anterior module long lens adapter with low magnification, to observe the limbal structure (POV). The purpose of the study is to assess the role of aging and regions on the limbus.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer control without ocular surface disease or prior ophthalmic surgery history

Exclusion Criteria:

* Patients who decline to receive the diagnostic examinations.
* Patients younger than 6 years old or older than 90 years old.

Ages: 6 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy normal eyes without any ocular surface disease
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
thickness of limbus | 1 day of inclusion
  measure the thickness of limbus from the image of OCT, describe the morphology of limbus (typical pattern was defined as having the easily identified sharp tapering tip of subepithelial stroma pointing to the corneal-limbal junction with the maximum epithelial thickness of palisades of Vogt at least 1.5 X thicker than the central corneal epithelial thickness)

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Li Chen, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan